CLINICAL TRIAL: NCT06609668
Title: Pilot Study to evaluateThrombomodulin to Rule Out Giant Cell Arteritis (GCA) in Polymyalgia Rheumatica (PMR) Patients. (THROPIQ)
Acronym: THROPIQ
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: RAMON AOI 2022
Record Dates: First submitted 2024-09-12; First posted 2024-09-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Giant Cell Arteritis (GCA); Polymyalgia Rheumatica (PMR)
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Additional blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Isolated PMR: 2012 PMR classification criteria GCA ACR/EULAR 2022 score < 6
  GCA ACR/EULAR 2022 score:
  * Shoulder/cervical spine pain/stiffness (+2)
  * Sudden loss of vision (+3)
  * Jaw claudication (+2)
  * Temporal headache (recent) (+2)
  * Scalp tenderness (+2)
  * Temporal artery abnormality on clinical examination (+2)
  * ESR > 50 mm/h or CRP > 10 mg/L (+3)
  * Positive TAB or halo sign (ultrasound) (+5)
  * Axillary artery involvement (+2)
  * Aortitis (hypermetabolism of the aorta) on FDG-PET (+2)
  Interventions: Biological: Additional blood samples
- PPR associated with GCA: * 2012 PMR classification criteria
  * ACR/EULAR 2022 score ≥ 6
  GCA ACR/EULAR 2022 score:
  * Shoulder/cervical spine pain/stiffness (+2)
  * Sudden loss of vision (+3)
  * Jaw claudication (+2)
  * Temporal headache (recent) (+2)
  * Scalp tenderness (+2)
  * Temporal artery abnormality on clinical examination (+2)
  * ESR > 50 mm/h or CRP > 10 mg/L (+3)
  * Positive TAB or halo sign (ultrasound) (+5)
  * Axillary artery involvement (+2)
  * Aortitis (hypermetabolism of the aorta) on FDG-PET (+2)
  Interventions: Biological: Additional blood samples

INTERVENTIONS:
Biological: Additional blood samples — * 1 dry tube (5 mL)
  * 1 EDTA tube (6 mL)
  Performed at inclusion (before any glucocorticoid and/or immunosuppressive treatment) and at follow-up visit (3 months after inclusion)

SUMMARY:
Polymyalgia rheumatica (PMR) is a rheumatologic condition occurring in patients > 50 years old, characterized by inflammatory pain of the scapular (shoulder) and pelvic (hip) girdles. PMR is most often isolated but can be associated with giant cell arteritis (GCA), a large vessels vasculitis, in 16 to 21% of case. The main features of GCA are headaches, jaw claudication, visual disturbances, abnormal temporal artery, scalp tenderness associated to elevated CRP and/or ESR. However, GCA could be asymptomatic in particular in case of isolated involvement of large vessels (subclinical GCA).

GCA requires high doses of glucocorticoids, compared to isolated PMR, to avoid complications resulting from vascular remodeling (stroke, blindness). Ruling out GCA in PMR patients relies on the performance of some complementary exams that explore cranial vessels as color doppler ultrasound and/or temporal artery biopsy and large vessels that relies on PET/FDG or angio CT scan.

The aim of this study is to identifie serum biomarkers that could rule out or identifies GCA in patients with PMR features. Ultimately, if biomarkers are identified, this could allow to select PMR patients in whom complementary exams are needed or not. For this study, investigators chose to explore thrombomodulin. Thrombomodulin is a protein that is increased in the circulating blood during vascular inflammation, and therefore seems to be a good candidate for distinguish isolated PMR from PMR associated with GCA.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given oral consent
* Patient > 50 years of age

Patients with PPR, meeting ACR/EULAR 2012 criteria:

* age > 50 years at onset of symptoms
* inflammatory limb-girdle pain
* elevated ESR (>20 mm/hr) and/or CRP (> 10 mg/l)
* AND Score ≥ 4 points among

  * Morning stiffness > 45 minutes (2 pts)
  * Hip pain or limitation of amplitude (1 pt)
  * Rheumatoid factor or anti-CCP antibodies negative (2 pts)
  * Absence of other joint pain (1 pt)

Exclusion Criteria:

* Patient not affiliated to national health insurance
* Patient under legal protection (curatorship, guardianship)
* Patient subject to a measure of legal safeguard
* Pregnant or breast-feeding women
* Adult patient unable to provide consent
* Patient having received corticosteroid or immunosuppressive treatment in the month prior to inclusion
* Patient with a contraindication to corticosteroid therapy
* Patients with an active infection, neoplasia or other inflammatory/autoimmune condition
* Patients with late onset rheumatoid arthritis.
* Conditions rendering vascular imaging unfeasible or uninterpretable:
* For angio-CT: allergy to iodine, renal failure (CKD <30 mL/min)
* For PET scan: unbalanced diabetes NB: only one of the two vascular imaging techniques will be performed, depending on the patient's condition and the technical resources available.

Secondary exclusion criteria:

* Final diagnosis of paraneoplastic PMR
* Final diagnosis of RA
* Negative PET scan (if performed 72 hours after glucocorticoid introduction)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Polymyalgia rheumatica (PMR)
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum thrombomodulin concentrations by Luminex at diagnosis (prior to any glucocorticoid treatment) | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France